CLINICAL TRIAL: NCT05619224
Title: Efficacy of a Physiotherapy Intervention to Improve Feeding Skills in Preterm Infants
Brief Title: Physiotherapy to Improve Feeding Skills in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, María del Mar Sánchez Joya, Associate Professor, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FiPrem
Record Dates: First submitted 2022-10-22; First posted 2022-11-16 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Premature Birth; Parenteral Nutrition; Motor Disorders; Neurodevelopmental Disorders; Sucking Behavior
Keywords: Premature Birth; Neurodevelopmental Disorders; NICU; Physical Stimulation
MeSH Terms: conditions — Premature Birth; Hyperphagia; Motor Disorders; Neurodevelopmental Disorders; Sucking Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GEO+N (Experimental): Neurodevelopmental stimulation intervention programme combined with an oral stimulation programme. They recives 10 sesions of 15 minutes of stimulation.
  Interventions: Other: Neurodevelopmental stimulation + Oral stimulation; Other: Oral stimulation
- GEO (Experimental): Oral stimulation programme. They recives 10 sesions of 15 minutes of stimulation.
  Interventions: Other: Oral stimulation

INTERVENTIONS:
Other: Neurodevelopmental stimulation + Oral stimulation — Neurodevelopmental intervention seeks to reduce abnormal postures and movement patterns in premature infants, allowing them to experience physiological postures in flexion and receive sensory stimulation. To this is added oral stimulation.
  These stimulations are performed on alternate days.
  Arms: GEO+N
Other: Oral stimulation — This intervention consists of performing a sensorimotor stimulation of oral structures: stimulating for 7 minutes perioral structures( cheeks, lips and jaw)intraoral structures for 5 minutes and in the last 3 minutes non-nutritive suction stimulation with pacifier or finger.

SUMMARY:
INTRODUCTION: Suction problems are very common in premature children due to a lack of maturation and orofacial control, the manifestation of a low muscle tone and the incoordination during sucking-swallow-breathe. In addition, there are some problems in different systems that get it worse.

AIM: compare oral stimulation programme with a neurodevelopmental stimulation intervention programme combined with an oral stimulation programme, evaluating its effectiveness on feeding development, neuromotor development and other aspects of development.

METHODOLOGY: we proposed a prospective parallel group clinical trial with two randomized and independent experimental groups. All preterm infants born between 2022-2023 at University Hospital Torrecárdenas, with nasogastric tube and gestational age between 27-32 weeks will be included.

EXPECTED BENEFITS: to have better results when the preterm infant is approached globally, also considering the postural situation of the preterm infant. In addition, it is expected that the development of children treated by combining oral stimulation with neurodevelopmental stimulation will be equated or close to healthy and born-to-term child.

RESULTS APPLICABILITY: Improved eating performances will reduce length of hospital stay as well as a greater autonomy improving family situation. It will also allow the reduction of hospital costs and the creation of a new way to attend this problem in preterm children.

ELIGIBILITY:
Inclusion Criteria:

Premature infants with a gestational age between 27 and 32 weeks, with an adequate weight for their gestational age, admitted to the unit of Neonatology, hemodynamically stable and with enteral nutrition

Exclusion Criteria:

* Neurological disorders
* Invasive mechanical ventilation
* Congenital disorders
* Necrotising enterocolitis
* Metabolic diseases
* Intraventricular hemorrhage grade 3-4
* Genetic disorders
* Oral disorders that make this process difficult(cleft palate, cleft lip...)
* Serious illnesses according to medical criteria

Ages: 27 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Transition time | Two years
  The transition time from tube to oral feeding. To complete this, the baby has to feed independently during two consecutive days.

SECONDARY OUTCOMES:
Feeding evolution | Two years
  Total oral amount
OFEATINg (Oral FEeding Assessment in premaTure Infants) | Two years
  To assess the ability for oral feeding. This scale was developed in two phases, the first phase being the design and construction of its items, and the second phase consisted of the analysis of the reliability and validity of this scale to through a cross-sectional study conducted in 2016/2017.
  The Oral FEeding Assessment in premaTure Infants may help clinicians to evaluate oral feeding readiness and oral feeding success, defned as the infant's ability to maintain physiologic stability (Alonso-Fernandez et al., 2022) The total score of the OFEATINg scale is the sum of the scores of all the items, with a minimum score of 13 and a maximum of 52, with a higher score reflecting greater readiness for oral feeding.
Weight | Two years
  With a scale in grames
Height | Two years
  With a measuring tape in millimeters.
Head circumference. | Two years
  With a measuring tape in millimeters.
PERI | Two years
  With the hospital discharge report we will be able to carry out the perinatal risk inventory (PERI) obtaining a numerical value that estimates the level of biological risk of the baby.
  Considering: low risk in scores from 0 to 6, moderate from 7 to 9 and high 10 or more.
  (Scheiner et al,. 1991)
Gross Motor Skills | Two years.
  In order to assess the quality of gross motor skills in the motor development of the baby we use the AIMS scale (Alberta Infant Motor Scale). The AIMS is an observational scale created by Canadian researchers to assess the motor development of children from birth to the acquisition of walking. Contains 58 items that assess the integrity and control of the antigravity muscles during different motor skills in prone position, supine position, sitting and standing(de Albuquerque et al, 2015).
Neuromotor Development | Two years
  To know the motor development and cognitive development and language.
  The Bayley ScaleIII scale is the most used tool to assess development, its main objective is to identify children with a developmental delay and provide information for plan of intervention. It is composed of 6 scales that allow assessing at the level of the cognitive, linguistic, motor, social-emotional, adaptive, and behavior of children between 1 and 42 months (de Albuquerque et al, 2018).
  With this scale we can determine the percentile the child has in each area of development, with a higher score reflects greater capabilities.
Neuromotor Development | Two years
  With the observation and analysis of the General Movements, you can get a lot of information about the situation of the child, allowing prognostic data to be provided to health professionals and family. The main objective of the GM's is to detect early the appearance of abnormal movements and predict possible cerebral palsy (Seesahai et al., 2021).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Torrecardenas, Almería, Almería, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available for one year once the study is finished
Access Criteria: Reasonable request to reproduce the intervention performed on this study

REFERENCES:
- [Background] Scheiner AP, Sexton ME. Prediction of developmental outcome using a perinatal risk inventory. Pediatrics. 1991 Dec;88(6):1135-43. PMID 1720234
- [Background] Alonso-Fernandez S, de Liria CRG, Lluch-Canut T, Poch-Pla L, Perapoch-Lopez J, Juve-Udina ME, Martinez-Momblan MA, Hurtado-Pardos B, Roldan-Merino JF. Psychometric properties of the oral feeding assessment in premature infants scale. Sci Rep. 2022 May 12;12(1):7836. doi: 10.1038/s41598-022-11521-0. PMID 35551222
- [Background] de Albuquerque PL, Lemos A, Guerra MQ, Eickmann SH. Accuracy of the Alberta Infant Motor Scale (AIMS) to detect developmental delay of gross motor skills in preterm infants: a systematic review. Dev Neurorehabil. 2015 Feb;18(1):15-21. doi: 10.3109/17518423.2014.955213. Epub 2014 Oct 3. PMID 25279804
- [Background] Albuquerque PL, Guerra MQF, Lima MC, Eickmann SH. Concurrent validity of the Alberta Infant Motor Scale to detect delayed gross motor development in preterm infants: A comparative study with the Bayley III. Dev Neurorehabil. 2018 Aug;21(6):408-414. doi: 10.1080/17518423.2017.1323974. Epub 2017 May 24. PMID 28537470
- [Background] Seesahai J, Luther M, Church PT, Maddalena P, Asztalos E, Rotter T, Banihani R. The assessment of general movements in term and late-preterm infants diagnosed with neonatal encephalopathy, as a predictive tool of cerebral palsy by 2 years of age-a scoping review. Syst Rev. 2021 Aug 12;10(1):226. doi: 10.1186/s13643-021-01765-8. PMID 34384482